CLINICAL TRIAL: NCT06427941
Title: A Phase 1 Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-B2033, Alone or in Combination With Tislelizumab With or Without Bevacizumab, in Participants With Selected Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 Study of BGB-B2033, Alone or in Combination With Tislelizumab With or Without Bevacizumab, in Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-B2033-101; 2025-524136-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hepatocellular Carcinoma; Local Advanced Hepatocellular Carcinoma; Alpha-fetoprotein (AFP)-Producing Gastric Cancer; Extragonadal Yolk Sac Tumors; Glypican-3 (GPC3)-Positive Squamous Non-small Cell Lung Cancer
Keywords: GPC-3; GPC3-positive squamous non-small cell lung cancer; BGB-B2033; tislelizumab; hepatocellular carcinoma; alpha-fetoprotein (AFP)-producing gastric cancer; extragonadal yolk sac tumors; Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular; Simpson-Golabi-Behmel syndrome | interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Monotherapy Dose Escalation and Safety Expansion) (Experimental): Ascending dose levels of BGB-B2033 monotherapy
  Interventions: Drug: BGB-B2033
- Part B (Combination Dose Escalation and Safety Expansion) (Experimental): Cohorts of BGB-B2033 in combination with tislelizumab
  Interventions: Drug: BGB-B2033; Drug: Tislelizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: BGB-B2033 — Administered by intravenous infusion
Drug: Tislelizumab — Administered by intravenous infusion
  Arms: Part B (Combination Dose Escalation and Safety Expansion)
Drug: Bevacizumab — Administered by intravenous infusion
  Arms: Part B (Combination Dose Escalation and Safety Expansion)

SUMMARY:
This is a first-in-human (FIH) clinical study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and anti-tumor activity of BGB-B2033 administered as monotherapy and in combination with tislelizumab, with or without bevacizumab. The study will enroll participants with locally advanced or metastatic hepatocellular carcinoma (HCC), alpha-fetoprotein (AFP)-producing gastric cancer (GC), extragonadal yolk sac tumors/non-dysgerminomas, or glypican-3 (GPC3)-positive squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must have one of the following unresectable, locally advanced, or metastatic tumor types:

   1. Hepatocellular carcinoma (HCC): Histologically or cytologically confirmed HCC that is either Barcelona Clinic Liver Cancer (BCLC) Stage C, or BCLC Stage B that is not amenable to, or has progressed after, loco-regional therapy and is not eligible for a curative treatment approach.
   2. Alpha-fetoprotein (AFP)-producing gastric cancer (GC): Histologically confirmed GC with AFP > 20 ng/mL in blood or tumor tissue positive for AFP by a validated immunohistochemistry (IHC) assay based on local or central testing.
   3. Germ cell tumors: Histologically confirmed germ cell tumors including extragonadal yolk sac tumors (e.g., located in the mediastinum, vagina, brain, retroperitoneum), and non-dysgerminomas for which no further curative systemic treatment options exist.
   4. Glypican-3 (GPC3)-positive squamous non-small cell lung cancer (NSCLC): Histologically confirmed GPC3-positive squamous NSCLC with prior exposure to a checkpoint inhibitor (CPI).
2. At least one evaluable lesion for dose escalation, and
3. At least one measurable lesion for safety expansion, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
5. Adequate organ function as defined in the protocol.
6. Provision of tumor tissue samples is required for specified parts of the study.

Key Exclusion Criteria:

1. Prior therapy directed against glypican-3 (GPC3) or the T-cell costimulatory receptor 4-1BB (CD137).
2. Active leptomeningeal disease or uncontrolled/untreated brain metastases.
3. Active autoimmune disease or a history of autoimmune disease with potential for relapse.
4. Any malignancy diagnosed ≤ 2 years before the first dose of study drug(s), except: The cancer type under investigation in this study, or Locally recurring malignancies previously treated with curative intent.
5. Requirement for systemic corticosteroids (> 10 mg/day prednisone or equivalent) or other immunosuppressive therapy within 14 days prior to the first dose of study drug(s).
6. Certain comorbidities involving the lungs, heart, bleeding conditions, or active infections, as defined in the protocol.

Note: Additional protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 2 years
  Number of participants with AEs and SAEs characterized by type, frequency, severity (as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5.0 [NCI-CTCAE v 5.0/American Society for Transplantation and Cellular Therapy [ASTCT] for cytokine release syndrome [CRS] and immune effector cell-associated neurotoxicity syndrome [ICANS]), timing, seriousness, and relationship to study therapy; assessment of adverse events meeting protocol-defined dose-limiting toxicity (DLT) criteria;
Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-B2033 | Up to approximately 2 years
  The MTD or MAD is defined as the highest dose that is tolerable or the highest dose administered, respectively.
Recommended Phase 2 dose (RP2D) of BGB-B2033 | Up to approximately 2 years
  The RP2D(s) will be determined based on a biologically effective dose by taking the totality of available preclinical and clinical data, including safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and antitumor activity, into consideration

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) using Response Evaluations Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease as determined from tumor assessments using RECIST v1.1.
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease using RECIST v1.1 or death, whichever occurs first.
Serum concentration of of BGB-B2033 | Up to approximately 2 years
Number of participants with anti-drug antibodies (ADAs) to BGB-B2033 | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (16):
- United States (3):
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Upmc Hillman Cancer Center(Univ of Pittsburgh), Pittsburgh, Pennsylvania
  - Scri Oncology Partners, Nashville, Tennessee
- China (9):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang Universityhongjiaozhou Branch, Nanchang, Jiangxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Auckland City Hospital, Auckland, New Zealand
- South Korea (3):
  - Cha Bundang Medical Center, Cha University, BundangGu SeongnamSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials